CLINICAL TRIAL: NCT06512259
Title: A Retrospective Study To Evaluate The Safety And Effectiveness Of AlloMend® Acellular Dermal Matrix Used In Post Mastectomy Pre-Pectoral Breast Reconstruction And Followed For Up To 6-Months Post-Operatively.
Brief Title: AlloMend Acellular Dermal Matrix Allograft in Pre-Pectoral Breast Reconstruction
Status: Recruiting | Type: Observational
Sponsor: AlloSource (Industry)
Responsible Party: Sponsor
Other Study IDs: ADM2023-001
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pre-Pectoral Breast Reconstruction Following Single or Double Mastectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AlloMend® Acellular Dermal Matrix allograft — AlloSource, a non-profit supplier of allografts and one of the nation's leading tissue banks, introduced AlloMend® Acellular Dermal Matrix allograft to bring the benefits of regenerative medicine to more patients. cellular allograft matrices, unlike synthetic materials or xenografts, are recognized as human tissue by the body for graft incorporation by the recipient, minimizing the risk of inflammation or rejection. AlloMend® Acellular Dermal Matrix allograft has been shown to incorporate into the surgical site and demonstrates blood vessel infiltration.

SUMMARY:
This is a single-center, retrospective study which will be used to describe and evaluate the effectiveness of AlloMend® Acellular Dermal Matrix allograft for patients that have undergone Pre-Pectoral Breast Reconstruction surgery following a single or double mastectomy.

DETAILED DESCRIPTION:
AlloMend® Acellular Dermal Matrix is a sterile, ready to use, human-derived acellular dermal matrix (ADM) allograft that can be used in a number of reconstructive and other surgical procedures. It is made from donated human full-thickness skin. After the epidermal and hypodermal layers are removed, the tissue is treated by a proprietary cleansing process.

AlloMend® is intended to be used in conjunction with a breast implant or tissue expander to stabilize implant position and minimize implant loss during post-single or double mastectomy, unilateral or bilateral pre-pectoral breast reconstruction in women 18 years of age or older. AlloMend® may be used in either one-stage (direct-to-implant) or two-stage (expander-to-implant) procedures.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following inclusion criteria to participate in this study:

* Diagnosed by a physician and required a single or double mastectomy followed by Pre-Pectoral Breast Reconstruction surgery with the use of AlloMend® Acellular Dermal Matrix allograft;
* Surgical intervention using AlloMend® Acellular Dermal Matrix allograft was used;
* Has completed or will complete the anticipated clinically indicated follow-up visits at 2 weeks, 6 weeks, 3 months, and 6 months post-surgical intervention.

Exclusion Criteria:

Patients must not meet any of the following criteria to be considered for this clinical trial:

* Did not utilize AlloMend® Acellular Dermal Matrix allograft during pre-pectoral breast reconstruction
* Did not have post-operative evaluations at the clinical site.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — AlloMend® is intended to be used in conjunction with a breast implant or tissue expander to stabilize implant position and minimize implant loss during post-single or double mastectomy, unilateral or bilateral pre-pectoral breast reconstruction in women 18 years of age or older. AlloMend® may be used in either one-stage (direct-to-implant) or two-stage (expander-to-implant) procedures.
Study Population: All patients who require a single or double mastectomy and have undergone a Pre-Pectoral Breast Reconstruction surgery with the use of AlloMend® Acellular Dermal Matrix allograft are eligible to participate. Patients who meet all of the inclusion criteria but do not meet any of the exclusion criteria are eligible to enter the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Descriptive Data Collection | Up to 6- months post-operatively
  The primary objective is to obtain descriptive data and surgical intervention and post operative surgical outcome data on AlloMend® Acellular Dermal Matrix allograft for patients that have undergone Pre-Pectoral Breast Reconstruction surgery following a single or double mastectomy.

SECONDARY OUTCOMES:
Physical Function and Quality of Life | Up to 6- months post-operatively
  Secondary Objectives will identify changes in physical function and quality of life as assessed for a period of 6-months post-operatively.

OTHER OUTCOMES:
Qualitative Data | Up to 6- months post-operatively
  Qualitative data such as return to wound healing, pain, discomfort, physicial deformity, and revision surgeries will also be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Alan H. Chen Surgical Associates, PC, Joliet, Illinois, United States